CLINICAL TRIAL: NCT01150474
Title: Randomized Clinical Trial of Postoperative Belladonna and Morphine Suppositories in Vaginal Surgery
Brief Title: Postoperative Belladonna and Morphine Suppositories in Vaginal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kristina A. Butler (Other)
Responsible Party: Sponsor-Investigator, Kristina A. Butler, M.D., Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-008045
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Vaginal Surgery
Keywords: Belladonna; Morphine; Suppositories; Vaginal; Surgery; Postoperative; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belladonna and Opium Suppositories (Experimental): Belladonna (16.2 mg) and opium (60 mg) suppositories administered rectally immediately following surgery and every 8 hours for 16 hours for a total of 3 doses.
  Interventions: Drug: Belladonna and Opium Suppositories
- Placebo Suppositories (Placebo Comparator): Placebo suppositories administered rectally immediately following surgery and every 8 hours for 16 hours for a total of 3 doses.
  Interventions: Drug: Placebo Suppositories

INTERVENTIONS:
Drug: Belladonna and Opium Suppositories — Belladonna (16.2 mg) and opium (60 mg) suppositories administered rectally immediately following surgery and every 8 hours for 16 hours for a total of 3 doses.
  Other Names: B & O Supprettes
  Arms: Belladonna and Opium Suppositories
Drug: Placebo Suppositories — Placebo suppositories administered rectally immediately following surgery and every 8 hours for 16 hours for a total of 3 doses.
  Arms: Placebo Suppositories

SUMMARY:
Our primary aim is to determine whether the routine use of belladonna and morphine suppositories will improve pain control following vaginal surgery. Treatment will begin immediately following surgery and every 8 hours for 16 hours.

DETAILED DESCRIPTION:
Minimizing postoperative pain is vital to a successful surgical recovery. Inadequate pain control may result in nausea, vomiting, an extended hospital stay, and reduced patient satisfaction. Oral and parenteral narcotics are commonly used for pain relief and their use may exacerbate the incidence of sedation, nausea, and vomiting; ultimately delaying convalescence. Previous studies have demonstrated that rectal analgesia following surgery results in lower pain scores and less intravenous morphine consumption. Belladonna and opium suppositories are routinely prescribed at our institution and their efficacy has not been confirmed.

A prospective, randomized, double-blind, placebo-controlled trial will be undertaken using belladonna and opium rectal suppositories following vaginal surgery. Treatment will begin immediately following surgery and continue every 8 hours for a total of 3 doses.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective vaginal surgery requiring general anesthesia at the Mayo Clinic Hospital. This would include a vaginal hysterectomy with culdoplasty or post-hysterectomy prolapse repair, including culdoplasty with or without anterior/posterior repair.

Exclusion Criteria:

* Participation in another trial using an investigational product.
* Pregnancy.
* Scheduled for a non-vaginal surgical procedure.
* Scheduled for a robotic hysterectomy.
* Scheduled to have combined surgeries (vaginal surgery plus another non-vaginal surgery).
* There is a known hypersensitivity to belladonna and/or opium.
* Contraindication to narcotic use.
* Chronic pain with preoperative pain score greater than 4 out of 10 points.
* Clinically significant substance abuse.
* Mental condition that may impair the ability to provide study assessments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Butler, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Mayo Clinic in Arizona, United States from January 2011 to April 2013.
Period: Overall Study
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Started | 51 | 52
Completed | 41 | 49
Not Completed | 10 | 3
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Cancer found | 1 | 0
Not completed — Multiple Studies | 0 | 1
Not completed — Rectotomy | 1 | 0
Not completed — Drug did not arrive in time | 1 | 0
Not completed — Drug not administered | 1 | 0
Not completed — Surgery Changed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories | Total
Number analyzed (Participants) | 41 | 49 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (12) | 55 (13) | 55 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 49 | 90
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 49 | 90
Pelvic Organ Prolapse [Number; unit: participants]
  Prolapse | 21 | 25 | 46
  No Prolapse | 20 | 24 | 44
Procedure time [Mean (Standard Deviation); unit: minutes] | 98 (37) | 96 (38) | 97 (37)
Estimated Blood Loss [Mean (Standard Deviation); unit: mL] | 180 (250) | 150 (110) | 161 (186)
Preoperative Pain [Mean (Standard Deviation); unit: units on a scale] — Pain was recorded on a validated numeric pain scale (1-10), with 0 = no pain and 10 = worst pain imaginable. Not all participants completed the pain scale, therefore the populations analyzed were Belladonna and Morphine Suppository Arm (N=39), Placebo Suppository Arm (N=45).
  units on a scale | 0.44 (1.25) | 0.24 (0.91) | 0.3 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Pain at Hour 4
Description: Pain at 4 hours was recorded using a linear analog pain scale, with 0 being "no pain," and 10 being "worst pain imaginable."
Time Frame: 4 hours following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Number analyzed (Participants) | 41 | 49
units on a scale | 4.2 (2.4) | 4.1 (2.1)
Statistical Analysis 1: Comparison: Belladonna and Opium Suppositories vs Placebo Suppositories; Test type: Superiority or Other; p = 0.82, t-test, 2 sided

2. Secondary Outcome: Pain at Hour 12
Description: Pain at 12 hours was recorded using a linear analog pain scale, with 0 being "no pain," and 10 being "worst pain imaginable."
Time Frame: 12 hours after surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Number analyzed (Participants) | 41 | 49
units on a scale | 3.4 (2.4) | 3.3 (2.2)
Statistical Analysis 1: Comparison: Belladonna and Opium Suppositories vs Placebo Suppositories; Test type: Superiority or Other; p = 0.75, t-test, 2 sided

3. Secondary Outcome: Pain at Hour 20
Description: Pain at 20 hours was recorded using a linear analog pain scale, with 0 being "no pain," and 10 being "worst pain imaginable."
Time Frame: 20 hours after surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Number analyzed (Participants) | 41 | 49
units on a scale | 2.5 (1.9) | 3.4 (2.5)
Statistical Analysis 1: Comparison: Belladonna and Opium Suppositories vs Placebo Suppositories; Test type: Superiority or Other; p = 0.07, t-test, 2 sided

4. Secondary Outcome: Narcotic Rescue Medication
Description: Use of all ancillary narcotic medications was taken from the medical record.
Time Frame: For 24 hours following surgery
Measure: Mean (Standard Deviation); unit: mg IV morphine equivalents
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Number analyzed (Participants) | 41 | 49
mg IV morphine equivalents | 57 (38) | 66 (61)
Statistical Analysis 1: Comparison: Belladonna and Opium Suppositories vs Placebo Suppositories; Test type: Superiority or Other; p = 0.43, t-test, 2 sided

5. Secondary Outcome: Number of Subjects With Nausea
Description: This information was taken from the medical record.
Time Frame: Approximately 12 hours after surgery
Measure: Number; unit: participants
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Number analyzed (Participants) | 41 | 49
participants | 14 | 22
Statistical Analysis 1: Comparison: Belladonna and Opium Suppositories vs Placebo Suppositories; Test type: Superiority or Other; p = 0.30, t-test, 2 sided

6. Secondary Outcome: Number of Subjects With Vomiting
Description: This information was taken from the medical record.
Time Frame: Within 20 hours of surgery
Measure: Number; unit: participants
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Number analyzed (Participants) | 41 | 49
participants | 13 | 9
Statistical Analysis 1: Comparison: Belladonna and Opium Suppositories vs Placebo Suppositories; Test type: Superiority or Other; p = 0.14, t-test, 2 sided

7. Secondary Outcome: Number of Times Antiemetic Rescue Medication Was Used
Time Frame: First 24 hours after surgery
Measure: Mean (Standard Deviation); unit: number of times antiemetics used
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Number analyzed (Participants) | 41 | 49
number of times antiemetics used | 1.7 (1.6) | 1.6 (1.5)
Statistical Analysis 1: Comparison: Belladonna and Opium Suppositories vs Placebo Suppositories; Test type: Superiority or Other; p = 0.83, t-test, 2 sided

8. Secondary Outcome: Number of Subjects Who Used Antiemetic Rescue Medications
Time Frame: First 24 hours after surgery
Measure: Number; unit: participants
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Number analyzed (Participants) | 41 | 49
participants | 30 | 33
Statistical Analysis 1: Comparison: Belladonna and Opium Suppositories vs Placebo Suppositories; Test type: Superiority or Other; p = 0.55, t-test, 2 sided

9. Secondary Outcome: Satisfaction With Pain Relief
Description: Patient satisfaction with pain relief was evaluated 24 hours after surgery using a linear analog satisfaction scale, with 0 being "very dissatisfied," and 10 being "very satisfied."
Time Frame: Approximately 24 hours following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Number analyzed (Participants) | 41 | 49
units on a scale | 8.2 (2.5) | 7.9 (2.6)
Statistical Analysis 1: Comparison: Belladonna and Opium Suppositories vs Placebo Suppositories; Test type: Superiority or Other; p = 0.59, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Subjects will be followed for 24 hours after surgery, and the research coordinator will assess for adverse events one week after surgery via the electronic medical record.
Arm/Group | Belladonna and Opium Suppositories | Placebo Suppositories
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/49
Other Adverse Events (participants affected / at risk) | 24/41 | 27/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belladonna and Opium Suppositories (N=41) | Placebo Suppositories (N=49)
Abdominal Sepsis (General disorders) | 1 (1) | 0 (0) — Within 24 hours of surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Belladonna and Opium Suppositories (N=41) | Placebo Suppositories (N=49)
Anemia Postoperative (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — Within 24 hours of surgery
Urinary Retention (Renal and urinary disorders) | 21 (21) | 23 (23) — Within 24 hours of surgery
Postoperative Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) — Within 24 hours of surgery
Procedural Hypertension (Cardiac disorders) | 1 (1) | 0 (0) — Within 24 hours of surgery
Pruritis Generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Within 24 hours of surgery
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — Within 24 hours of surgery
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Within 24 hours of surgery
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Within 24 hours of surgery
Procedural Hypotension (Cardiac disorders) | 1 (1) | 3 (3) — Within 24 hours of surgery
Constipation (Gastrointestinal disorders) | 20/35 (20) | 27/46 (27) — Within 7 days of surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes